CLINICAL TRIAL: NCT00769847
Title: Endoscopic Treatment for Isolated, Single Suture Craniosynostosis
Status: Withdrawn | Type: Observational
Why Stopped: Study was withdrawn due to lack of resources.
Sponsor: University of Utah (Other)
Responsible Party: Faizi Siddiqi, M.D., Principal Investigator, University of Utah
Other Study IDs: 22034
Record Dates: First submitted 2008-10-07; First posted 2008-10-09 (Estimated); Last update posted 2015-06-02 (Estimated); Status verified 2015-05

CONDITIONS: Craniosynostosis
Keywords: Endoscopic, craniosynostosis, sagittal, synostosis
MeSH Terms: conditions — Craniosynostoses; Synostosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Sagittal synostosis: Male and female infants from 1-6 months of age with isolated, single suture sagittal craniosynostosis.
  Interventions: Procedure: Endoscopic strip craniectomy

INTERVENTIONS:
Procedure: Endoscopic strip craniectomy — Surgery

SUMMARY:
This is a prospective study to evaluate outcomes in patients undergoing endoscopic craniectomy for isolated, single-suture craniosynostosis.

ELIGIBILITY:
Inclusion Criteria:

* Infants 1 to 6 months of age with isolated, single-suture craniosynostosis.

Exclusion Criteria:

* Multiple suture craniosynostosis and infants older than 6 months of age.

Ages: 1 Month to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Male and female infants, from 1 to 6 months of age with isolated, single-suture sagittal craniosynostosis.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-09; Primary Completion 2009-07 (Actual); Study Completion 2013-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Faizi Siddiqu, MD, Principal Investigator — University of Utah

REFERENCES:
- [Background] Obrien MO, Johnson M: Craniosynostosis, in Youmans JR (ed): Neurological Surgery, Philadelphia: WB Saunders, 1990, Vol 2, p 1328.
- [Background] HAAS LL. Roentgenological skull measurements and their diagnostic applications. Am J Roentgenol Radium Ther Nucl Med. 1952 Feb;67(2):197-209. No abstract available. PMID 14903268
- [Background] Lannelongue M. De la craniectomie dans la microcephalie. Compt Rend Seances Acad Sci 50:1382-1385, 1890.
- [Background] Lane LC. Pioneer craniectomy for the relief of mental imbecility due to premature sutural closure and microcephalus. JAMA 18:49-50, 1892.
- [Background] Panchal J, Marsh JL, Park TS, Kaufman B, Pilgram T, Huang SH. Sagittal craniosynostosis outcome assessment for two methods and timings of intervention. Plast Reconstr Surg. 1999 May;103(6):1574-84. doi: 10.1097/00006534-199905060-00004. PMID 10323690
- [Background] Jimenez DF, Barone CM. Endoscopic craniectomy for early surgical correction of sagittal craniosynostosis. J Neurosurg. 1998 Jan;88(1):77-81. doi: 10.3171/jns.1998.88.1.0077. PMID 9420076
- [Background] Jimenez DF, Barone CM, McGee ME, Cartwright CC, Baker CL. Endoscopy-assisted wide-vertex craniectomy, barrel stave osteotomies, and postoperative helmet molding therapy in the management of sagittal suture craniosynostosis. J Neurosurg. 2004 May;100(5 Suppl Pediatrics):407-17. doi: 10.3171/ped.2004.100.5.0407. PMID 15287447
- [Background] Murad GJ, Clayman M, Seagle MB, White S, Perkins LA, Pincus DW. Endoscopic-assisted repair of craniosynostosis. Neurosurg Focus. 2005 Dec 15;19(6):E6. doi: 10.3171/foc.2005.19.6.7. PMID 16398483